CLINICAL TRIAL: NCT04054128
Title: Bicarbonate vs Heparin Catheter Lock in Chronic Hemodialysis Patients
Acronym: BICATH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital General "Dr. Miguel Silva" de Morelia (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); NAUSLIFE HEMODIALYSIS CLINICS (Unknown)
Responsible Party: Principal Investigator, J ARMANDO VÁZQUEZ ÁVILA, MD, Nephrology fellow, Hospital General "Dr. Miguel Silva" de Morelia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 479/01/19
Record Dates: First submitted 2019-07-23; First posted 2019-08-13 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: End Stage Renal Disease; Vascular Access Complication; Catheter Complications; Hemodialysis Access Failure; Hemodialysis Catheter Infection
Keywords: Sodium bicarbonate lock; Heparin lock; Vascular access complication
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Sodium Bicarbonate; Injections; Heparin

STUDY DESIGN:
Intervention Model Description: Prospective, open label, clinical trial in chronic hemodialysis patients with a catheter as a vascular access, randomized to bicarbonate lock or heparin lock (control) as standard treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium bicarbonate catheter lock group (SBCL) (Experimental): Chronic hemodialysis patients with a catheter as a vascular access, will be lock with sodium bicarbonate 7.5% Injection.
  Interventions: Drug: Sodium Bicarbonate 7.5% Injection
- Heparin catheter lock group (HCL) (Active Comparator): Chronic hemodialysis patients with a catheter as a vascular access, will be lock with heparin, 1000 Units/mL injectable solution
  Interventions: Drug: Heparin Sodium, 1000 Units/mL Injectable Solution 1

INTERVENTIONS:
Drug: Sodium Bicarbonate 7.5% Injection — Sodium bicarbonate solution for catheter lock; 7.5% sodium bicarbonate solution will be used for catheter lock in both catheter lumens, 1.9 mL in each catheter lumen will be infused after hemodialysis treatment during 3 months.
  Other Names: Bicarnat® arm
  Arms: Sodium bicarbonate catheter lock group (SBCL)
Drug: Heparin Sodium, 1000 Units/mL Injectable Solution 1 — Heparin for catheter lock: 1000 u/mL heparin solution will be used for catheter lock in both catheter lumens as standard treatment, 1.9 mL in each catheter lumen will be infused after hemodialysis treatment during 3 months.
  Other Names: Inhepar® arm
  Arms: Heparin catheter lock group (HCL)

SUMMARY:
Prospective clinical trial to evaluate the efficacy of catheter lock with bicarbonate vs heparin in chronic hemodialysis patients. Two groups will be created, sodium bicarbonate lock group (experimental group) and heparin lock group (control group). Catheter pressures, flow, patency and infection outcomes will be compare between groups at different time points (30, 60 and 90 days).

DETAILED DESCRIPTION:
A prospective, randomized, clinical, open-label trial at Hospital General "Dr. Miguel Silva" de Morelia, Mexico.

The study period will be between august 16, 2019 to November 16, 2019. The aim of this study is to evaluate the efficacy of catheter lock with bicarbonate vs heparin in chronic hemodialysis patients. Primary outcome will be catheter function. Secondary outcomes will be Infectious complications, thrombotic complications, and frequency of adverse effects between groups.

All patients provided written informed consent before enrollment. The trial protocol was approved by Hospital General "Dr. Miguel Silva" Internal Review Board, register number 17-CI-16053153, and Research & Ethics committee, with register number 16-CEI-004-20161212, Study registry # 479/01/9.

Patients between 18-65 years old, incident or prevalent chronic hemodialysis, with 1 month of clinical stability and with temporal catheter as vascular access for hemodialysis are eligible. A total of 60 patients will be included in the study. All patients will be randomly assigned into one of two groups: SBCL (n=30), intervention group and HCL (n=30), as control group.

Before each hemodialysis treatment, catheters and connections will be inspected for leaks, evidence of damage, exit-site infection and tunnel infection. Intraluminal SBCL or HCL solution will be removed before connecting the hemodialysis catheter to a dialysis machine prior to any treatment.

During each treatment, patients will be prescribed and monitored for complications and standard treatment will be provided to every patient. After each treatment, blood will be rinsed from dialysis lines with 0.9% saline solution back to the patient. Upon the conclusion of treatment, all catheters will be flushed with 10 mL 0.9% saline solution per blood line respectively, after saline flush, catheter lock will be prescribed; SBCL group with 7.5% sodium bicarbonate solution, at a dose of 2 milliliters per lumen, and HCL group with sodium heparin at a concentration of 1000 units per milliliter, at a dose of 2 milliliters per lumen. Catheter exit site dressing changes occurred after each HD treatment.

Niagra 13.5 French/20 cm non tunneled catheter will be the standard vascular access. All central venous catheters will be inserted by an expert operator under strict aseptic protocol. Catheter care will be performed by trained dialysis staff. At the end of dialysis, all catheters will be flushed and locked with the respectively arm solution.

Function assessment will be based on both, pressure and flow measurements on arterial line, as well as measurements of arterial and venous line pressures and flow during hemodialysis sessions. Infectious and thrombotic complications will be assessed as defined.

ELIGIBILITY:
Inclusion Criteria:

* Patients who accept participation and sign informed consent.
* Incident or prevalent chronic hemodialysis patients who receive at least 2 sessions per week with 1 month of clinical stability defined as: no hospitalizations, no vascular access infections, no changes in blood flow prescription due to vascular access dysfunction.
* Patients with temporal catheter (Niagra 13.5 French/20 cm length, BARD Access System, Salt Lake City, Utah, USA) as vascular access for hemodialysis.

Exclusion Criteria:

* Catheter dysfunction at baseline
* On anticoagulation therapy
* Patients with known coagulopathy or hemophilia
* Patients with Child-Pugh B or C liver failure
* Patients with thrombocytopenia less than 100,000 u / L
* Patients with central vessel stenosis and vena cava syndrome, previously documented.
* Patients with vascular access exhaustion.
* Patients who have undergone more than 2 vascular approaches for hemodialysis catheters.
* Patients with heparin-induced thrombocytopenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-09-28 (Estimated)

PRIMARY OUTCOMES:
Arterial line pressure at fixed blood flow in sodium bicarbonate lock versus heparin lock catheters in chronic hemodialysis patients | 30 days.
  Arterial line pressure[mmHg] at 300 mL/min blood flow will be compared between sodium bicarbonate lock and heparin lock in chronic hemodialysis patients.
Arterial line pressure at fixed blood flow in sodium bicarbonate lock versus heparin lock catheters in chronic hemodialysis patients | 60 days
  Arterial line pressure[mmHg] at 300 mL/min blood flow will be compared between sodium bicarbonate lock and heparin lock in chronic hemodialysis patients.
Arterial line pressure at fixed blood flow in sodium bicarbonate lock versus heparin lock catheters in chronic hemodialysis patients | 90 days
  Arterial line pressure[mmHg] at 300 mL/min blood flow will be compared between sodium bicarbonate lock and heparin lock in chronic hemodialysis patients.

SECONDARY OUTCOMES:
Incidence rate of catheter related bloodstream infection | 90 days
  Catheter related bloodstream infection rate (events per 100 days/catheter) will be compare between sodium bicarbonate lock versus heparin lock in chronic hemodialysis patients
Incidence rate of catheter thrombosis | 90 days
  Catheter thrombosis rate (events per 100 days/catheter) will be compare between sodium bicarbonate lock versus heparin lock in chronic hemodialysis patients
Adverse events incidence | 90 days
  To compare the frequency of hemorrhagic event, anaphylaxis, hypernatremia or death between sodium bicarbonate lock vs heparin lock in chronic hemodialysis patients

CONTACTS AND LOCATIONS:
Overall Officials: Israel Campos, M.D., Principal Investigator — Hospital General "Dr. Miguel Silva" de Morelia
Locations (1):
- Hospital General "Dr. Miguel Silva" de Morelia, Morelia, Michoacán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jha V, Garcia-Garcia G, Iseki K, Li Z, Naicker S, Plattner B, Saran R, Wang AY, Yang CW. Chronic kidney disease: global dimension and perspectives. Lancet. 2013 Jul 20;382(9888):260-72. doi: 10.1016/S0140-6736(13)60687-X. Epub 2013 May 31. PMID 23727169
- [Background] Ma A, Shroff R, Hothi D, Lopez MM, Veligratli F, Calder F, Rees L. A comparison of arteriovenous fistulas and central venous lines for long-term chronic haemodialysis. Pediatr Nephrol. 2013 Feb;28(2):321-6. doi: 10.1007/s00467-012-2318-2. Epub 2012 Oct 6. PMID 23052655
- [Background] Adib-Hajbaghery M, Molavizadeh N, Alavi NM. Quality of care of vascular access in hemodialysis patients in a hemodialysis center in Iran. J Vasc Nurs. 2012 Mar;30(1):24-8. doi: 10.1016/j.jvn.2011.10.002. PMID 22321404
- [Background] Agharazii M, Plamondon I, Lebel M, Douville P, Desmeules S. Estimation of heparin leak into the systemic circulation after central venous catheter heparin lock. Nephrol Dial Transplant. 2005 Jun;20(6):1238-40. doi: 10.1093/ndt/gfh841. Epub 2005 Apr 26. PMID 15855206
- [Background] Moran JE, Ash SR; ASDIN Clinical Practice Committee. Locking solutions for hemodialysis catheters; heparin and citrate--a position paper by ASDIN. Semin Dial. 2008 Sep-Oct;21(5):490-2. doi: 10.1111/j.1525-139X.2008.00466.x. Epub 2008 Aug 29. PMID 18764795
- [Background] Chen FK, Li JJ, Song Y, Zhang YY, Chen P, Zhao CZ, Gong HY, Yao DF. Concentrated sodium chloride catheter lock solution--a new effective alternative method for hemodialysis patients with high bleeding risk. Ren Fail. 2014 Feb;36(1):17-22. doi: 10.3109/0886022X.2013.830207. Epub 2013 Sep 2. PMID 23992231
- [Background] Palomo I, Pereira J, Alarcon M, Diaz G, Hidalgo P, Pizarro I, Jara E, Rojas P, Quiroga G, Moore-Carrasco R. Prevalence of heparin-induced antibodies in patients with chronic renal failure undergoing hemodialysis. J Clin Lab Anal. 2005;19(5):189-95. doi: 10.1002/jcla.20076. PMID 16170812
- [Background] Yon CK, Low CL. Sodium citrate 4% versus heparin as a lock solution in hemodialysis patients with central venous catheters. Am J Health Syst Pharm. 2013 Jan 15;70(2):131-6. doi: 10.2146/ajhp120300. PMID 23292266
- [Background] Shanks RM, Sargent JL, Martinez RM, Graber ML, O'Toole GA. Catheter lock solutions influence staphylococcal biofilm formation on abiotic surfaces. Nephrol Dial Transplant. 2006 Aug;21(8):2247-55. doi: 10.1093/ndt/gfl170. Epub 2006 Apr 20. PMID 16627606
- [Background] Zhao Y, Li Z, Zhang L, Yang J, Yang Y, Tang Y, Fu P. Citrate versus heparin lock for hemodialysis catheters: a systematic review and meta-analysis of randomized controlled trials. Am J Kidney Dis. 2014 Mar;63(3):479-90. doi: 10.1053/j.ajkd.2013.08.016. Epub 2013 Oct 11. PMID 24125729
- [Background] Beigi AA, HadiZadeh MS, Salimi F, Ghaheri H. Heparin compared with normal saline to maintain patency of permanent double lumen hemodialysis catheters: A randomized controlled trial. Adv Biomed Res. 2014 May 28;3:121. doi: 10.4103/2277-9175.133192. eCollection 2014. PMID 24949292
- [Background] Zhong L, Wang HL, Xu B, Yuan Y, Wang X, Zhang YY, Ji L, Pan ZM, Hu ZS. Normal saline versus heparin for patency of central venous catheters in adult patients - a systematic review and meta-analysis. Crit Care. 2017 Jan 8;21(1):5. doi: 10.1186/s13054-016-1585-x. PMID 28063456
- [Background] Wong DW, Mishkin FS, Tanaka TT. The effects of bicarbonate on blood coagulation. JAMA. 1980 Jul 4;244(1):61-2. PMID 7382058
- [Background] Farha MA, French S, Stokes JM, Brown ED. Bicarbonate Alters Bacterial Susceptibility to Antibiotics by Targeting the Proton Motive Force. ACS Infect Dis. 2018 Mar 9;4(3):382-390. doi: 10.1021/acsinfecdis.7b00194. Epub 2018 Jan 4. PMID 29264917
- [Background] Nostro A, Cellini L, Di Giulio M, D'Arrigo M, Marino A, Blanco AR, Favaloro A, Cutroneo G, Bisignano G. Effect of alkaline pH on staphylococcal biofilm formation. APMIS. 2012 Sep;120(9):733-42. doi: 10.1111/j.1600-0463.2012.02900.x. Epub 2012 Apr 11. PMID 22882263